CLINICAL TRIAL: NCT00192296
Title: A Phase I, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability,Immunogenicity, and Pharmacokinetics of MEDI-528, a Humanized Monoclonal Anti-Interleukin-9 Antibody, in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability,Immunogenicity, and Pharmacokinetics of MEDI-528 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP105
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — enokizumab

ARMS (4):
- MEDI-528 0.3 mg/kg (Experimental): MEDI-528 (0.3 mg/kg) administered as a single, intravenous (IV) dose
  Interventions: Biological: MEDI-528 0.3 mg/kg
- MEDI-528 1 mg/kg (Experimental): MEDI-528 (1 mg/kg) administered as a single, IV dose
  Interventions: Biological: MEDI-528 1 mg/kg
- MEDI-528 3 mg/kg (Experimental): MEDI-528 (3 mg/kg) administered as a single, IV dose
  Interventions: Biological: MEDI-528 3 mg/kg
- MEDI-528 9 mg/kg (Experimental): MEDI-528 (9 mg/kg) administered as a single, IV dose
  Interventions: Biological: MEDI-528 9 mg/kg

INTERVENTIONS:
Biological: MEDI-528 0.3 mg/kg — MEDI-528 (0.3 mg/kg) administered as a single, intravenous (IV) dose
  Arms: MEDI-528 0.3 mg/kg
Biological: MEDI-528 1 mg/kg — MEDI-528 (1 mg/kg) administered as a single, IV dose
  Arms: MEDI-528 1 mg/kg
Biological: MEDI-528 3 mg/kg — MEDI-528 (3 mg/kg) administered as a single, IV dose
  Arms: MEDI-528 3 mg/kg
Biological: MEDI-528 9 mg/kg — MEDI-528 (9 mg/kg) administered as a single, IV dose
  Arms: MEDI-528 9 mg/kg

SUMMARY:
Phase I study to evaluate the safety and tolerability of escalating single IV doses of MEDI-528.

DETAILED DESCRIPTION:
The primary objective of this Phase I study is to evaluate the safety and tolerability of escalating single IV doses of MEDI-528 administered to healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 up to and including 49 years of age at the time of the first dose of study drug
* Weight < 89 kg
* Written informed consent obtained from the volunteer
* Healthy by medical history and physical examination
* Sexually active females, unless surgically sterile or at least one year post-menopausal, must use an effective method of avoiding pregnancy (including oral, injectable, transdermal or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap,abstinence, use of a condom by the sexual partner or sterile sexual partner) for 3 months before the first dose of study drug, and must agree to continue using such precautions through 84 days after their dose of study drug. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active males, unless surgically sterile, must likewise use an effective method of birth control (condom or abstinence) and must agree to continue using such precautions through 84 days after their dose of study drug.
* Use of common over-the-counter medications such as topical corticosteroids, decongestants, antihistamines, analgesics, and antacids is permitted unless, in the opinion of the investigator, it would interfere with either the volunteer's ability to complete the study or interpretation of study results.
* Ability to complete the follow-up period of 84 days
* Willing to forego other forms of experimental treatment during the study period of 84 days

Exclusion Criteria:

* Acute illnesses or evidence of significant active infection, such as fever ≥38.0°C (100.5°F) at the start of the study
* Use of prescription medications, other than contraceptives, in the 28-day period before Study Day 0
* Blood donation in excess of 400 mL within 6 months of the time of entry into the study
* History of use of tobacco products within 3 years of Study Day 0 or history of smoking of >10 pack-years
* History of immunodeficiency or receipt or current use of immunosuppressive drugs including systemic corticosteroids
* History of allergic disease or reactions likely to be exacerbated by any component of the Study Drug (described in the Investigator's Brochure)
* History of substance abuse that, in the opinion of the investigator, may compromise the ability of the study subject to complete the study and follow-up period
* Evidence of any systemic disease on physical examination
* Evidence of infection with hepatitis A, B, or C virus or HIV-1
* Receipt of immunoglobulins or blood products within 60 days of entering the study
* Receipt of any investigational drug therapy within 60 days of the first dose of study drug through Study Day 84 (use of licensed agents for indications not listed in the package insert is permitted)
* Any of the following: CBC: Hgb < 12.0 gm/dL; WBC < 4,000/mm3; platelet count <125,000/mm3 (or laboratory normal values); Na, K, Cl, CO2, AST, ALT, BUN, 4-hour fasting glucose, amylase, lipase, creatinine, troponin > upper limit of normal; other abnormal laboratory values in the screening panel which in the opinion of the principal investigator are judged to be clinically significant.
* Clinically significant abnormality, as determined by the investigator, on 12-lead electrocardiogram at the time of initial screening
* Elective surgery planned during the study period through Study Day 84
* Pregnancy (sexually active females must have a negative serum pregnancy test on the day of the first dose of the study drug, before dosing)
* Nursing mother
* The presence of any acute or chronic organ-specific condition or any concern, which in the opinion of the investigator, may interfere with the conduct or interpretation of the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-08; Primary Completion 2005-02 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Vargas, MD, Principal Investigator
Locations (1):
- MDS Pharma Services, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] White B, Leon F, White W, Robbie G. Two first-in-human, open-label, phase I dose-escalation safety trials of MEDI-528, a monoclonal antibody against interleukin-9, in healthy adult volunteers. Clin Ther. 2009 Apr;31(4):728-40. doi: 10.1016/j.clinthera.2009.04.019. PMID 19446146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants provided written informed consent and participated in the study between 13Aug2004 and 12Nov2004 at one site in New Orleans, Louisiana.
Pre-assignment Details: Eligible participants received MEDI-528 in an open-label manner.
Period: Overall Study
Arm/Group | MEDI-528 0.3 mg | MEDI-528 1 mg | MEDI-528 3 mg | MEDI-528 9 mg
Started | 6 | 6 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI-528 0.3 mg | MEDI-528 1 mg | MEDI-528 3 mg | MEDI-528 9 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.8 (11.1) | 29.8 (8.4) | 25.5 (8.8) | 30.5 (8.2) | 27.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 4 | 4 | 13
  Male | 6 | 1 | 2 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Number of participants experiencing adverse events (includes both adverse events and serious adverse events)
Time Frame: Days 0 - 84
Population: All subjects who received MEDI-528
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 5 | 4 | 6 | 2

2. Primary Outcome: Incidence of Abnormal Troponin Levels
Description: Number of participants with troponin levels greater than upper limit of normal (> 0.05 ng/mL)
Time Frame: Days 0, 7, 14, 21, and 28
Population: All subjects who received MEDI-528
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of Serious Adverse Events
Description: Number of participants experiencing serious adverse events
Time Frame: Days 0 - 84
Population: All subjects who received MEDI-528
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) to MEDI-528
Description: Number of participants who had ADA detected at each time point
Time Frame: Days 14, 28, 42, and 84
Population: All subjects who received MEDI-528
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Day 14 | 0 | 0 | 0 | 0
  Day 28 | 0 | 0 | 0 | 0
  Day 42 | 0 | 0 | 0 | 0
  Day 84 | 0 | 0 | 1 | 0

5. Secondary Outcome: Time to Observed Maximum Serum Concentration (Tmax)
Description: Tmax of MEDI-528
Time Frame: Days 0 (prior to and after the end of the infusion, and at 1, 2, 4, 8, and 12 hours after the end of the infusion), 1, 3, 5, 7, 10, 14, 21, 28, 42, and 84
Population: All subjects who received MEDI-528
Measure: Median (Full Range); unit: Hours
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours | 1.5 (0.0) [0.0 to 4.0] | 1.1 [0.1 to 2.1] | 1.2 [0.2 to 24.2] | 0.7 [0.5 to 2.6]

6. Secondary Outcome: Observed Maximum Serum Concentration (Cmax)
Description: Cmax of MEDI-528
Time Frame: as for outcome 5
Population: All subjects who received MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Micrograms per milliliter | 7.2 (42) | 22.2 (30) | 59.7 (25) | 231.2 (17)

7. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Last Measurable Concentration [AUC(0-t)]
Description: AUC(0-t) of MEDI-528
Time Frame: as for outcome 5
Population: All subjects who received MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms times hours per milliliter
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Micrograms times hours per milliliter | 2463.7 (85) | 7765.6 (55) | 26221.5 (40) | 101476.7 (16)

8. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Infinity [AUC(0-infinity)]
Description: AUC(0-infinity) of MEDI-528
Time Frame: as for outcome 5
Population: All subjects who received MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram times hours per milliliter
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Microgram times hours per milliliter | 3982.2 (67) | 10084.6 (50) | 30035.5 (40) | 112344.3 (22)

9. Secondary Outcome: Percent of Total Area Under the Concentration Curve Extrapolated From Last Measurable Time to Infinity [AUC(Ext)]
Description: AUC(ext) of MEDI-528
Time Frame: as for outcome 5
Population: All subjects who received MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Projected AUC
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of Projected AUC | 35.8 (30) | 21.5 (30) | 10.5 (64) | 8.2 (63)

10. Secondary Outcome: Total Body Clearance (CL)
Description: CL of MEDI-528
Time Frame: Days 0, 1, 3, 5, 7, 10, 14, 21, 28, 42, and 84
Population: All subjects who received MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliter per day
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Milliter per day | 120.5 (51) | 160.1 (34) | 166.1 (31) | 154.6 (13)

11. Secondary Outcome: Half-life (T1/2)
Description: T1/2 of MEDI-528
Time Frame: Days 0, 1, 3, 5, 7, 10, 14, 21, 28, 42, and 84
Population: All subjects who received MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours | 651.1 (24) | 559.1 (36) | 581.3 (21) | 594.9 (26)

12. Secondary Outcome: Terminal Phase Elimination Rate (Vz)
Description: Vz of MEDI-528
Time Frame: Days 0, 1, 3, 5, 7, 10, 14, 21, 28, 42, and 84
Population: All subjects who received MEDI-528
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liters | 4.7 (38) | 5.4 (30) | 5.8 (19) | 5.5 (18)

ADVERSE EVENTS:
Time Frame: Days 0-84
Arm/Group | MEDI-528 0.3 mg | MEDI-528 1 mg | MEDI-528 3 mg | MEDI-528 9 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 6/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-528 0.3 mg (N=6) | MEDI-528 1 mg (N=6) | MEDI-528 3 mg (N=6) | MEDI-528 9 mg (N=6)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
White blood cell count decreased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.